CLINICAL TRIAL: NCT05816291
Title: A Randomized, Crossover Pilot to Examine the Acute Impact of Veillonella Supplementation on Exercise and Lactate Responses
Brief Title: Pilot Study to Examine the Acute Impact of Veillonella Supplementation on Exercise and Lactate Responses
Acronym: VP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Collaborators: Increnovo, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-22-60
Record Dates: First submitted 2023-03-14; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Lactate Blood Increase; Exhaustion - Physiological
Keywords: Blood Lactate; Physiological Exhaustion; Exercise
MeSH Terms: conditions — Hyperlactatemia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to ingest one of two supplement conditions in a randomized, double-blind, and crossover fashion. A randomized order of treatments will be generated by random.org.
Who Masked: Participant, Investigator
Masking Description: The same number of capsules will be provided to each participant. Each capsule will be identical in color, shape, smell, and transparency. Participants will be instructed to consume their assigned dose with 8 - 12 fluid ounces of cool water.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 14 days of supplementation placebo (maltodextrin)
  Interventions: Dietary Supplement: Time to Exhaustion at velocity at VO2max
- Veillonella atypica FB004 (Experimental): 14 days of supplementation 1 x 109CFU dose Veillonella atypica FB004
  Interventions: Dietary Supplement: Time to Exhaustion at velocity at VO2max

INTERVENTIONS:
Dietary Supplement: Time to Exhaustion at velocity at VO2max — During a familiarization trial prior to supplementation and before and after each supplementation period at the beginning of each study visit, participants will complete a standardized warm-up consisting of walking on a treadmill for 5 minutes, a series of whole-body dynamic movements (high knees, butt kicks, walking lunges, straight-leg marching, etc.), and a self-prescribed period of jogging on the treadmill for no more than ten minutes. The speed on the treadmill will then be set at the velocity upon which 100% VO2Peak was achieved. Participants will be instructed to run at this velocity for as long as they can. No feedback in terms of duration, pacing, etc. will be provided, and participants will be provided verbal encouragement to run for as long as possible.
  Other Names: TTW

SUMMARY:
The purpose of this study is to assess the health and performance outcomes associated with supplementation of Veillonella atypica.

DETAILED DESCRIPTION:
This pilot study will be conducted using a randomized, double-blind, crossover study design. Healthy men and women (n=7) between the ages of 18 - 50 years of age will be recruited for this study. After signing an IRB-approved consent form, participants will have their peak VO2 determined to finalize eligibility. Eligible participants will then practice their first time to exhaustion trial at 100% VO2Peak. Prior to each subsequent study visit, participants will be scheduled at a similar time between the hours of 0600 and 1000 hours and will be asked to observe an overnight fast (food, caffeine, and nicotine) while refraining from any vigorous exercise for at least 24 hours prior to their visit. During visit 2, participants will have their body composition assessed and complete another time to exhaustion familiarization at 100% VO2Peak. Leading up to and during each subsequent study visit (identical to visit 3), participants will collect a stool sample and upon arrival at the laboratory have their body mass measured before having a venous blood sample collected for assessment of complete blood count and comprehensive metabolic panel. After blood collection, participants will complete the standardized warm-up before completing a treadmill time to exhaustion test at 100% VO2Peak. Capillary lactate levels will be assessed before, immediately after, and 5 minutes after completion of the exhaustion trial using a handheld lactate analyzer. From there and in a randomized, double-blind, placebo-controlled, crossover fashion, participants will be assigned for the next 14 days to ingest either a placebo (maltodextrin) or a 1 x 109CFU dose of Veillonella atypica FB004 (VA) (Fitbiomics, Inc. New York). After supplementing for 14 days, participants will complete an identical battery of tests. Participants will then follow a wash-out period for 21 days before returning to the laboratory to complete study visit 5, the pre-supplementation visit to their supplementation period. After completing study visit 5, participants will be instructed to supplement with the alternative supplement for 14 days before returning for a 6th and final study visit. Participants will complete a two-day food and fluid record prior to visit 3, receivea copy of it from study investigators, and be instructed to replicate it prior to each subsequent study visit.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary signed and dated informed consent.
* Be in good health as determined by medical history and routine blood chemistries.
* Age between 18 and 50
* Exercises > 150 mins/week
* Body Mass Index of 18.5-29.9 and Body Fat of 30%
* Normotensive (seated, resting systolic blood pressure < 140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5 minute) rest period, and two more measurements will be taken. The average of all three measurements will be used to determine eligibility.
* Normal seated, resting heart rate (< 90 beats per minute). Willing to follow all study protocols.

Exclusion Criteria:

* Individuals currently diagnosed or being treated for any cardiac, respiratory, endocrine, psychiatric, musculoskeletal, renal, hepatic, neuromuscular or metabolic disease or disorder that in the judgement of the study participant's personal physician or research nurse that will preclude their safe participation or will contraindicate quality control over the collected data
* Individuals currently diagnosed with or are being treated for celiac disease, lactose intolerance, digestive insufficiencies or other gastrointestinal complications such as irritable bowel syndrome, ulcerative colitis, etc.
* Alcohol consumption (more than 2 standard alcoholic drinks per day or more than 10 drinks per week) or drug abuse or dependence.
* Smokers or individuals who have quit smoking within the last 6 months
* Known sensitivity to any ingredient in the test formulations as listed in the Nutrition Facts label.
* Individuals who are determined to be on a ketogenic diet.
* Individuals who are cognitively impaired and/or who are unable to give informed consent.
* Individuals taking a medication known to impact digestive function or hormonal functions that may impact how our body digests, absorbs, or metabolizes nutrients
* Individuals currently taking a probiotic or a dietary supplement that may impact digestive function or hormonal functions that may impact how our body digests, absorbs, or metabolizes nutrients
* Pregnant women, women trying to become pregnant, or nursing women.
* Participants who indicate they are actively restricting calories or attempting to lose weight.
* Individuals who do not participate in aerobic exercise > 2 days/week
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose a significant risk to the subject.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Aerobic Exercise Performance | 2 weeks
  Time to Exhaustion treadmill running at 100% VO2peak
Blood lactate response to intense exercise | 2 weeks
  Blood lactate response to treadmill running at 100% VO2peak protocol til exhaustion

SECONDARY OUTCOMES:
Alpha and beta diversity of veillonella atypica (fecal samples) | 2 weeks
  Alpha and beta diversity of veillonella atypica (fecal samples)
Changes in blood Hemoglobin concentration | 2 weeks
  Complete Blood Count (CBC) with Differential includes: Changes in blood Hemoglobin concentration
Changes in blood hematocrit | 2 weeks
  Complete Blood Count (CBC) with Differential includes: Changes in blood hematocrit
Changes in red blood cell count | 2 weeks
  Complete Blood Count (CBC) with Differential includes: Changes in red blood cell count
Changes in red blood cell distribution width | 2 weeks
  Complete Blood Count (CBC) with Differential includes: Changes in red blood cell distribution width
Changes in mean corpuscular volume (MCV) | 2 weeks
  Complete Blood Count (CBC) with Differential includes: Changes in mean corpuscular volume (MCV)
Changes in mean corpuscular hemoglobin concentration (MCHC) | 2 weeks
  Complete Blood Count (CBC) with Differential includes: Changes in mean corpuscular hemoglobin concentration (MCHC)
Changes in mean corpuscular hemoglobin (MCH) | 2 weeks
  Complete Blood Count (CBC) with Differential includes: Changes in mean corpuscular hemoglobin (MCH)
Changes in white blood cell count | 2 weeks
  Complete Blood Count (CBC) with Differential includes: Changes in white blood cell count
Changes in platelet count | 2 weeks
  Complete Blood Count (CBC) with Differential includes: Changes in platelet count
Changes in basophils | 2 weeks
  Complete Blood Count (CBC) with Differential includes: Changes in basophils
Changes in eosinophils | 2 weeks
  Complete Blood Count (CBC) with Differential includes: Changes in eosinophils
Changes in neutrophils | 2 weeks
  Complete Blood Count (CBC) with Differential includes: Changes in neutrophils
Changes in blood Glucose Concentration | 2 weeks
  Comprehensive metabolic Panel (CMP) includes: Changes in blood glucose Concentration
Changes in blood Sodium Concentration | 2 weeks
  Comprehensive metabolic Panel (CMP) includes: Changes in blood Sodium Concentration
Changes in blood Potassium Concentration | 2 weeks
  Comprehensive metabolic Panel (CMP) includes: Changes in blood Potassium Concentration
Changes in blood Chloride Concentration | 2 weeks
  Comprehensive metabolic Panel (CMP) includes: Changes in blood Chloride Concentration
Changes in blood Carbon Dioxide Concentration | 2 weeks
  Comprehensive metabolic Panel (CMP) includes: Changes in blood Carbon Dioxide Concentration
Changes in blood Calcium Concentration | 2 weeks
  Comprehensive metabolic Panel (CMP) includes: Changes in blood Calcium Concentration
Changes in blood alkaline phosphate Concentration | 2 weeks
  Comprehensive metabolic Panel (CMP) includes: Changes in blood alkaline phosphate Concentration
Changes in blood creatinine Concentration | 2 weeks
  Comprehensive metabolic Panel (CMP) includes: Changes in blood creatinine Concentration
Changes in blood Bilirubin Concentration | 2 weeks
  Comprehensive metabolic Panel (CMP) includes: Changes in blood Bilirubin Concentration
Changes in blood Blood Urea Nitrogen (BUN) Concentration | 2 weeks
  Comprehensive metabolic Panel (CMP) includes: Changes in blood Blood Urea Nitrogen (BUN) Concentration
Changes in blood Albumin Concentration | 2 weeks
  Comprehensive metabolic Panel (CMP) includes: Changes in blood Albumin Concentration
Changes in blood Globulin Concentration | 2 weeks
  Comprehensive metabolic Panel (CMP) includes: Changes in blood Globulin Concentration
Changes in blood total protein Concentration | 2 weeks
  Comprehensive metabolic Panel (CMP) includes: Changes in blood total protein Concentration
Changes in blood Aspartate aminotransferase (AST) Concentration | 2 weeks
  Comprehensive metabolic Panel (CMP) includes: Changes in blood Aspartate aminotransferase (AST) Concentration
Changes in blood Alanine Aminotransferase (ALT) Concentration | 2 weeks
  Comprehensive metabolic Panel (CMP) includes: Changes in blood Alanine Aminotransferase (ALT) Concentration

OTHER OUTCOMES:
Changes in Resting Heart Rate | 2 weeks
  Resting Heart Rate (beats per minute)
Changes in Systolic Blood Pressure | 2 weeks
  Changes in systolic blood pressure (mmHg)
Changes in Diastolic Blood Pressure | 2 weeks
  Changes in diastolic blood pressure (mmHg)
Occurrences of Reported adverse events | 2 weeks
  Occurrences of Reported adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise and Performance Nutrition Laboratory, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No